CLINICAL TRIAL: NCT03344263
Title: Study of the Reversibility of Vigilance Dysfunction at 6 Months of Continuous Positive Airways Pressure (CPAP) in Patients With Obstructive Sleep
Brief Title: Study of the Reversibility of Vigilance Dysfunction at 6 Months of Continuous Positive Airways Pressure (CPAP) in Patients With Obstructive Sleep Apnea/Hypopnea Syndrome (OSAHS)
Acronym: VISA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISA
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Vigilance Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tests of attentional performance (Experimental)
  Interventions: Diagnostic Test: tests of attentional performance

INTERVENTIONS:
Diagnostic Test: tests of attentional performance — tests of attentional performance before and after 6 months of continuous positive airways pressure

SUMMARY:
It is a monocentric prospective pilot study in Poitiers University Hospital, specifically analyzing the vigilance disorders in the Obstructive Sleep Apnea Hypopnea Syndrome (OSAHS) and their reversibility after 6 months of Continuous positive airways pressure (CPAP).

All subjects were administered a test of vigilance (Test of Attentional Performance) both before and after the 6 months of CPAP.

The main objective is the study of the reversibility of alertness disorders on the number of omissions in the subtest visual vigilance of the TAP ( (Test of Attentional Performance) at 6 months of CPAP in the OSAHS in patients with a memory complaint.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-70 years
* Memory disorders without memory problems in episodic memory
* Presence of polysomnography of a obstructive sleep apnea/hypopnea syndrome (OSAHS) requiring Continuous positive airways pressure

  * Moderate OSAHS (Apnea Hypopnea Index ≥ 15 / hour with arousals ≥ 10)
  * Severe OSAHS (Apnea Hypopnea Index ≥ 30 / h)

Exclusion Criteria:

* Age <20 years or ≥ 70 years
* Neurodegenerative disease (Alzheimer's disease, Parkinson's disease)
* Dysthyroidism
* Severe depression, schizophrenia, bipolar disorder
* Treatment with an effect on cognition: hypnotics, sedative
* Chronic Obstructive Pulmonary Disease
* Chronic alcoholism, other addictions
* Contraindications to Magnetic Resonance Imaging
* Refusal of equipment

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2021-02-09 (Actual); Study Completion 2021-02-09 (Actual)

PRIMARY OUTCOMES:
Study of the reversibility of vigilance disorders on the number of omissions in the subtest visual vigilance of the TAP | After 6 months of continuous positive airways pressure in the OSAHS patient
  Reversibility of vigilance disorders on the number of omissions in the subtest visual vigilance of the TAP

CONTACTS AND LOCATIONS:
Locations (1):
- service de neurologie CHU DE POITIERS, Poitiers, France